CLINICAL TRIAL: NCT02271737
Title: Newborn Infection Control and Care Initiative for Health Facilities to Accelerate Reduction of Newborn Mortality
Acronym: NICCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Institute of Public Health, Cambodia (Other Government)
Collaborators: Tulane University School of Public Health and Tropical Medicine (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Var Chivorn, Principle Investigator, National Institute of Public Health, Cambodia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15
Record Dates: First submitted 2014-10-05; First posted 2014-10-22 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Neonatal Infection
Keywords: Newborn; infection; community health
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Improve infection control in health centers; improve home hygiene; improve newborn danger signs recognition by the HC staff, VHSG, and mothers; and improve care coordination between community and health facilities. The above improvements will be through the training of health center staff and VHSG; HC staff and VHSG provide health education to mothers at the health centers and at home respectively; and provide supportive supervision to both HC and VHSG. VHSG will conduct three home visits to the mothers/newborns on the first 24 hours, the 3rd day, and the 7th day after delivery.
  Interventions: Behavioral: Training HC/VHSG, Health Education, and Supportive Supervision
- No Intervention (No Intervention): We do not make any interventions.

INTERVENTIONS:
Behavioral: Training HC/VHSG, Health Education, and Supportive Supervision — 1. Improve infection control Practice at health centers; 2) improve knowledge on newborn danger signs among HC staff, VHSG, and the mothers; 3) improve care coordination between community and health facilities, e.g. improve referral of sick newborns
  Arms: Experimental

SUMMARY:
Newborn mortality continues to be unacceptably high in Cambodia, despite reductions in maternal and under five year old mortality. Evidence exists that a large proportion of newborn mortality globally and in Cambodia is attributable to infections and sepsis. The study proposes a package intervention to address infection control in the perinatal period in facilities and to improve the timeliness of referral of newborns with suspected infections to appropriate health facilities for treatment through upgrading of hygiene practices in facilities and linking of community based volunteers with health facilities and families in the community setting.

By delivering a coordinated intervention that combines improved education for health center midwives, village health care workers, and mothers of newborns, along with improved care coordination with increase in number of interactions (points of contact) between mothers and health care personnel, the investigators will see improved knowledge of newborn danger signs among mothers and health care workers, more rapid case detection of significant newborn illnesses, and more rapid and appropriate referral of ill newborns.

The investigators also hypothesize that the common causes of newborn sepsis in Cambodia are different from those reported in Western cultures, and that Staphylococcus aureus will be a common pathogen as described in neighboring Laos. The investigators will evaluate the causes of newborn sepsis in the subset of infants referred to Takeo Provincial Hospital.

DETAILED DESCRIPTION:
The study will incorporate mixed methods: formative (qualitative) research, and a stepped wedge cluster randomized intervention trial and process evaluation. It is anticipated that the results of this study will provide data for policy level actions on newborn survival in Cambodia and in other settings with similar health outcomes. The study may contribute to the potential scale up of a linked model of community-facility care for newborns.

Globally, infection causes approximately 35% of all newborn mortality [1]. Verbal autopsy data collected in Svay Rieng province in 2009 show that bacterial sepsis is the likely cause in 40% of newborn deaths, by far the largest category (exceeding the next highest cause by 17%) [2].

The NICCI intervention addresses a number of barriers identified by the Royal Government of Cambodia and USAID to improving neonatal survival, including the capacity and performance of health providers to deliver newborn care through strengthened training; upgrading hygiene through enhanced infection control in facilities; and increasing community engagement in the demand for and delivery of health services for newborns through improving referral processes and addressing barriers to timely care seeking. The proposed study will address the crucial gap in post-natal care by linking the community (via Village Health Support Groups) with Health Center staff to follow mothers and newborns during the first week of life

Quality Assurance: Investigators will include provision for the management of all data collection and will include appropriate procedures in a Standard Operating Practices document. Training of data collectors at the start of the study will ensure quality and consistency and supervisory monitoring of data collection will occur monthly.

Data Checks and Data Source Verification: Data will be collected, checked, and entered into a data management system at the National Institute of Public Health. All participants will be identified by a unique identifier which will be the link for all databases. All study data will be collected by project staff so outcomes do not depend on subject compliance other than refusal to answer project surveys (although study participants always have a right to decline to answer a survey based on informed consent principles). Data collected in the community will be transferred to central databases at NIPH and entered into a database using REDcap or a comparable program that is compatible with data management capacity at NIPH. The investigators will use special screens with filters for invalid entries and identification of missing values for data entry verification. Analysis will be conducted in SPSS and/or SAS.

Sample Size: Using all cause newborn mortality as the primary outcome and stepped wedge design sample size calculation (power analysis) for cluster randomized trials, the investigators required a total sample size of 1,938 subjects based on 80% power, 5% significance level, and 10% rate of loss-to-follow up to detect a 20% reduction with a baseline neonatal mortality of 40 deaths/1,000 live births in target provinces and an intra-class correlation coefficient of 0.0007256.

Withdrawal from the Study: Study subjects may withdraw voluntarily from participation at any time. Participants may also voluntarily withdraw from receiving the study intervention at any time. The study team will attempt to follow those who withdraw from the study in order to collect safety data if applicable.

Termination of Study: Although very unlikely, discontinuation would occur if a statistically significant increase or decrease in neonatal deaths was detected in the intervention area and reasons for that correlated in any way to the content of the intervention.

Formative Study:

The investigators will conduct qualitative data collection from FGD with staff from 15 health centers, one-on-one interview with 20 VHSG and with 30 mothers of newborn. The study will allow us to get an overall knowledge on the knowledge and practices on newborn by HC and community before the implementation phase.

The baseline data will be collected from the comparison cluster during the course of intervention phase, environmental assessment checklist used in the health facilities which the investigators will use before the start of the intervention and during the interventions, and the planned formative research.

Intervention Study:

Determine the 1st HC for conducting the intervention. The investigators will randomly select one health center (HC) from among the 16 HCs. For the second and the subsequent HCs, the investigators will select the HC which is close to the first HC, and the investigators will continue this process until all the 16 HC are selected.

Training HC Staff: during the training for the first HC (which will be happening in the first month of the intervention phase), MCH (Maternal and Child Health) Focal Person and SC will conduct the training and HC Coordinators/other project staff will observe the training. Subsequent training for the HC staff will be conducted by HC Coordinators with the supervision support from Provincial Health Department (PHD) MCH Focal Person and SC. NICCI will conduct training for one HC each month. Before each training starts, the trainers will introduce a HC Data Form (only the relevant parts) to collect baseline data from the trainees. This training will go over a period of 16 months for the 16 health centers.

Training VHSG: during the first month of the intervention phase, the investigators will also organize training for VHSG under the HC's coverage (one HC at a time). This training will go over a period of 16 months. Before each training starts, the trainers will introduce VHSG Data Form (only relevant parts) to collect baseline data from the trainees.

Blood Samples from Sick Newborn: The investigators anticipate that pathogenic bacteria will be isolated in about 10% of the 200-300 blood samples to be tested over the 2 year period of the intervention-control study.

HC Coordinators Conduct Supportive Supervision to HC Staff in Intervention Clusters: the two HC Coordinators will jointly conduct monthly supportive supervision to the HC under the Invention Cluster. During the supervision, the HC Coordinators will perform the following:

Check whether NICCI's training/education materials for HC are available and used by HC staff; discuss with HC staff whether the staff recall 6 newborn danger signs and hygiene messages (hygiene for mothers/newborn/home and hygiene for HC staff themselves including knowledge on infection control); re-enforce HC staff (observe if applicable) to provide education to mothers on newborn care, newborn danger signs, and hygiene at home; re-enforce the practice of infection control according to NICCI training materials, and check whether HC staff have the skill and the materials/supplies to implement the infection control activities as written in the training materials; review birth register and ANC registers to assist HC staff in care coordination and assist VHSG Coordinators in pregnant women enrollment, e.g. HC communicate more effectively with VHSG; check whether HC staff, who provide ANC services, ask the pregnant women about meeting with VHSG in their villages, if the pregnant women have not met VHSG, HC needs to provide information about the pregnant women to relevant VHSG (call VHSG telephone), HC Coordinators can assist in this activity by comparing the name of pregnant women in the HC ANC register with the enrollment list; check whether the HC staff have done their work on care coordination with VHSG (e.g. call VHSG after the mother/newborn leave the HC) and inform VHSG on pregnant women enrollment as they have been trained; re-enforce this practice or confirm the HC staff if the HC staff have done properly; check whether the HC has an update enrollment list (so that HC staff know whether a woman come for delivery is the study participant). HC Coordinators need to work with VHSG Coordinators to ensure that HC staff have an up to date list (e.g. up to a month preceding the month in which HC Coordinator conduct the supervision).

The two HC Coordinators must have a supportive supervision book to record what activities the HC Coordinators have done during each supervision visit, with a clear supervision date and name of the HC. The record for each supervision visit should be ended by a summary of the finding and follow up actions.

HC Coordinators Conduct Weekly Visit to Each HC Under Comparison Clusters: the purpose of the visit is to collect information about the enrolled participants who have birth delivery in the HC so that the project has the information to interview the mothers/newborn in their villages on the 14th and 28th day after the delivery. In the visit, HC Coordinators collect the information and share the information with Data Manager. The Data Manager registers the information in the database and provide information to VHSG Coordinators for the VHSG Coordinators to meet each mother/newborn on the 14th day and on the 28th day. The information include: participant name and ID, and date of delivery. During the visit, HC Coordinators will also provide up to date enrollment list to the HC. It is also an option if the HC Coordinators think that they can secure this activity without visiting the HC and with only communicate with the HC through mobile phone

VHSG Coordinators Conduct Supportive Supervision to VHSG in Intervention Cluster: each VHSG Coordinator will be assigned to be responsible for approx. 54 villages, and needs to conduct supervision to each village every two months; the supervision will be conducted only for villages where VHSG have already been trained by NICCI. With the guidance from SC, VHSG Coordinators will develop a written schedule for VHSG supervision (two monthly schedule, which is equal to one round of supervision). During the supervision to each eligible village (meeting VHSG), the VHSG Coordinators will perform the following:

Check VHSG Pregnant Women Register to see whether VHSG has conducted proper registration: complete the register correctly, seem to register all the pregnant women (according to the estimated number of pregnant women in each village) Check VHSG whether they have communicated with their relevant HC on: mother coming home and other care coordination, and whether HC informed them about pregnant women in their villages and who have not been registered or contacted by the VHSG.

Discuss with VHSG about their knowledge, re-enforce their knowledge on: 6 newborn danger signs, newborn care as in the training/education materials, home hygiene by the family, message on care seeking; and check whether the VHSG have and use the NICCI's training/education/thermometer materials and re-enforce the use of the education materials when necessary.

Discuss whether VHSG conduct the three visits to mother/newborn: 24hours, 3rd, and 7th day, and discuss with VHSG whether they understand and use the VHSG Home Visit's materials.

Enroll/interview new pregnant women (using Consent Form and the Enrollment and Baseline Form), provide the completed forms to the Data Manager.

Each VHSG Coordinator must have a supervision record book, recording activities they have done during each supervision visit to each village (with name of VHSG), with a summary of the findings and clear follow up actions. SC will design this supervision Record Book for the VHSG Coordinators.

VHSG Coordinators Enroll Pregnant Women in Comparison Clusters: each VHSG Coordinator will travel to their designated villages under the comparison cluster every two months. During each visit, the VHSG Coordinators will perform the followings:

Discuss with VHSG to assist them in completing the pregnant women registration Meet with pregnant women (with the support from VHSG) who meet the criteria of enrollment (e.g. at their last semester of pregnancy) to enroll the pregnant women using Consent Form, and the Enrollment and Baseline Form.

HC Coordinators Conduct Data Collection from HC: the two HC Coordinators will jointly conduct the data collection from each HC every six months, using HC Data Collection Form. After completing, the HC Coordinators send the Form to Data Manager for his/her verification and data entry. SC and Data Manager will work closely with and assist HC Coordinators in the development of data collection plan for each data collection round (one round lasts for six month). The Data Manager will help SC to closely monitor HC Coordinators in adhering to the data collection plan and provide prompt feedback to SC and HC Coordinators.

VHSG Coordinators Conduct Data Collection from VHSG: each VHSG Coordinator will conduct interview with VHSG who work in their designated villages (approx. 50 village per VHSG Coordinator) every six month, using VHSG Data Form. After completing the Form, VHSG Coordinators send the completed Form to Data Manager for his/her verification and data entry. SC and Data Manager will work closely with and assist VHSG Coordinators in the development of data collection plan for each data collection round (one round lasts for six month), the Data Manager will help SC to closely monitor VHSG Coordinators in adhering to the data collection plan and provide prompt feedback to SC and VHSG Coordinators.

VHSG Coordinators Conduct Data Collection from Mothers/Caretakers: each VHSG Coordinator ensures that all registered mother/newborn (in his or her designated villages) are interviewed on the 14th and the 28th day after delivery. To know whether VHSG Coordinator has a mother/newborn to interview for a month, the VHSG Coordinator needs to work closely with the data manager who will generate the list of mother/newborn to visit on the 14th and on the 28th day.

ELIGIBILITY:
Inclusion Criteria:

* Health Centers: historically, a health center which providing services for more than 20 births per month
* Individuals: women in the last trimester of pregnancy with any ethnicity, age is equal or older than 18 years, and pregnancy results in a live birth.

Exclusion Criteria:

* Birth of baby with known congenital malformation
* Inability to obtain informed consent or adhere to protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1938 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
% of mothers who know at last 3 danger signs | 2 years
% of VHSG who know 6 danger signs | 2 years
% of families who seek care from an appropriate facility | 2 years
Time between onset of suspected danger signs and referral to appropriate facility | 2 years
Improved hygiene behavior by family | 2 years
  It is a composite score of: 1) % of mothers/caretakers interviewed said they wash hand after going to toilet; 2) % of mothers/caretakers interviewed said that they wash hand before touching newborn; 3) % of mothers/caretakers interviewed said that they wash hand before eating; and 4) % of mothers/caretakers interviewed said that they wash hand after cleaning baby's bottom.
Improved infection control behavior among HC staff | 2 years
  A composite score from: % of HC staff reported that they washed hands: 1) before patient contact (when they examine mother and newborn); 2) Before and after aseptic procedure; 3) After expose to blood/body fluids; 4) after patient contact (after removing gloves); and 5) after touching patient surroundings

SECONDARY OUTCOMES:
% of newborns visited at least once by VHSG on or before day 7 of life | 2 years
% of newborns visited at least twice by VHSG on or before day 7 of life | 2 years
% of VHSG who can deliver hygiene messages | 2 years
% of mothers who received messages on hygiene from HC staff | 2 years
% of mothers who received messages on hygiene from VHSG | 2 years
% of mothers who received messages on care seeking from VHSG | 2 years
% of HC staff who know 6 danger signs | 2 years
% of HC staff who recall hygiene messages | 2 years

OTHER OUTCOMES:
All causes newborn mortality | 2 years
Age and cause specific mortality rates | 2 years
Incidence rate of newborns with the following danger signs: convulsion, respiratory distress, fever or hypothermia, lethargy, and skin pustules | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Oberhelman Richard Alfred, MD, Study Chair — Tulane University; Alessandra N Bazzano, PhD, Study Chair — Tulane University; Chivorn Var, MD, MPH, Principal Investigator — National Institute of Public Heath, Cambodia; Navapol IvEk, MD, MPH, Study Director — National Institute of Public Health, Cambodia
Locations (1):
- Selected Health Centers and Villages Under the Health Centers, Takeo, Takeo Province, Cambodia

REFERENCES:
- [Background] National Maternal Child Health Center, Verbal Autopsy Study Svay Rieng, Ministry of Health, Editor 2009
- [Result] Lawn JE, Wilczynska-Ketende K, Cousens SN. Estimating the causes of 4 million neonatal deaths in the year 2000. Int J Epidemiol. 2006 Jun;35(3):706-18. doi: 10.1093/ije/dyl043. Epub 2006 Mar 23. PMID 16556647
- [Derived] Var C, Bazzano AN, Srivastav SK, Welty JC, Ek NI, Oberhelman RA. Newborn Infection Control and Care Initiative for health facilities to accelerate reduction of newborn mortality (NICCI): study protocol for a randomized controlled trial. Trials. 2015 Jun 5;16:257. doi: 10.1186/s13063-015-0771-5. PMID 26044715